CLINICAL TRIAL: NCT02180997
Title: Pharmacokinetic Drug Interaction Between Solifenacin 10mg and Tamsulosin 0.4mg in Healthy Male Volunteers
Brief Title: Clinical Trial to Investigate the Pharmacokinetic Drug Interaction Between Solifenacin and Tamsulosin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JLP-1207-P1-DI
Record Dates: First submitted 2014-07-01; First posted 2014-07-03 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2014-07

CONDITIONS: LUTS; Benign Prostatic Hyperplasia; Overactive Bladder
Keywords: α1-blockers; antimuscarinic agent
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Bladder, Overactive | interventions — Tamsulosin; Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Tamsulosin 1 (Experimental): Volunteers will be taken Tamsulosin and solifenacin
  Interventions: Drug: Solifenacin; Drug: Tamsulosin and solifenacin
- Solifenacin 1 (Experimental): Volunteers will be taken Tamsulosin and solifenacin
  Interventions: Drug: Tamsulosin; Drug: Tamsulosin and solifenacin
- Co-administration 1 (Experimental): Volunteers will be taken Tamsulosin and solifenacin
  Interventions: Drug: Tamsulosin; Drug: Solifenacin
- Tamsulosin 2 (Experimental): Volunteers will be taken Tamsulosin and solifenacin
  Interventions: Drug: Solifenacin; Drug: Tamsulosin and solifenacin
- Solifenacin 2 (Experimental): Volunteers will be taken Tamsulosin and solifenacin
  Interventions: Drug: Tamsulosin; Drug: Tamsulosin and solifenacin
- Co-administration 2 (Experimental): Volunteers will be taken Tamsulosin and solifenacin
  Interventions: Drug: Tamsulosin; Drug: Solifenacin

INTERVENTIONS:
Drug: Tamsulosin — Tamsulosin and solifenacin: Tamsulosin 0.4mg, once daily
  Other Names: Harnal-D tablet
  Arms: Co-administration 1; Co-administration 2; Solifenacin 1; Solifenacin 2
Drug: Solifenacin — Tamsulosin and solifenacin: Solifenacin 10 mg, once daily
  Other Names: Vesicare tablet
  Arms: Co-administration 1; Co-administration 2; Tamsulosin 1; Tamsulosin 2
Drug: Tamsulosin and solifenacin — Tamsulosin and solifenacin: Tamsulosin 0.4mg, once daily, Solifenacin 10 mg, once daily
  Other Names: Harnal-D and Vesicare tablet
  Arms: Solifenacin 1; Solifenacin 2; Tamsulosin 1; Tamsulosin 2

SUMMARY:
The purpose of this study is to investigate the pharmacokinetic drug interaction between Solifenacin and Tamsulosin in healthy male volunteers.

DETAILED DESCRIPTION:
Pharmacokinetic Drug Interaction Between Solifenacin 10mg and Tamsulosin 0.4mg in Healthy Male Volunteers

ELIGIBILITY:
Inclusion Criteria:

* 19~45 years healthy male
* Body weight is over 55kg, BMI measurement 18.0kg/m^2~ 27.0kg/m^2
* Signed informed consent form from to participate voluntarily and to comply with the trial requirements.
* Researchers determined suitable volunteers through physical examination, laboratory tests

Exclusion Criteria:

* History of clinically significant liver, kidneys, nervous system, immune system, respiratory, endocrine disorders or tumor or blood disorders, cardiovascular diseases, mental disorders (mood disorders, obsessive-compulsive disorder, etc.)
* Sitting SBP>150mmHg or <100mmHg, sitting DBP>100mmHg or <60mmHg, after 3 minutes break
* An impossible one who participants in clinical trial by investigator's decision including laboratory test result or another reason.
* Have a gastrointestinal disease history that can affect drug absorption (Crohn's disease ulcers, etc) or surgery (except simple appendectomy or hernia surgery)
* History of drug abuse
* Positive urine drug screening
* Administrated investigational product in a previous clinical trial within 90 days of the first administration day in this study.
* Donated blood within 60 days prior to the first administration day in this study.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss, Cmax,ss | 192h

SECONDARY OUTCOMES:
C trough,ss | 192h
Tmax,ss | 192h
t1/2 | 192h
CL/F | 192h

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-sang Yu, M.D.,Ph.D., Principal Investigator — Seoul National University Hospital(SNUH)
Locations (1):
- Seoul National University Hospital(SNUH), Seoul, Jongno-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No